CLINICAL TRIAL: NCT02445898
Title: Effect of Preoperative Intravenous High Dose Methylprednisolone on Orthostatic Intolerance and Heart Rate Variability in Patients Scheduled for Total Hip-arthroplasty
Brief Title: Effect of Methylprednisolone on Orthostatic Intolerance and Heart Rate Variability in Hip-arthroplasty Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Viktoria Oline Lindberg-Larsen, MD, PhD student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: HK_VL_01_2015; 2015-000102-19 (EudraCT Number)
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Osteoarthrosis
Keywords: Glucocorticoid; Orthostatic Intolerance; Heart Rate Variability; Hip arthroplasty, total
MeSH Terms: conditions — Osteoarthritis; Orthostatic Intolerance | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylprednisolone (Active Comparator): Preoperative single high dose of Solu-Medrol 125 mg iv.
  Interventions: Drug: Methylprednisolone
- Isotonic Sodium Chloride (Placebo Comparator): Preoperative single dose of isotonic Sodium Chloride
  Interventions: Drug: Isotonic Sodium Chloride

INTERVENTIONS:
Drug: Methylprednisolone — Comparison of preoperative single high dose of Methylprednisolone 125 mg iv. and isotonic Sodium Chloride (placebo)
  Other Names: Solu-Medrol
  Arms: Methylprednisolone
Drug: Isotonic Sodium Chloride — Placebo
  Arms: Isotonic Sodium Chloride

SUMMARY:
The study evaluates the pathophysiological effects of a single dose Methylprednisolone administered prior to total hip-arthroplasty (THA) surgery. The investigators examine the effect on orthostatic intolerance, orthostatic hypotension and heart rate variability (HRV) to evaluate the efficacy of Methylprednisolone regarding blood pressure regulation and autonomic responses after THA.

Half of participants will receive intravenous Solu-Medrol 125 mg, while the other half will receive placebo.

The investigators hypothesize that the group receiving Methylprednisolone will be less orthostatic intolerant, experience less orthostatic hypotension and have an improved autonomic response compared to the placebo-group, early after THA.

DETAILED DESCRIPTION:
The anti-inflammatory effects of glucocorticoids are well known. The beneficial effects in postoperative pain, postoperative nausea and vomiting are well-documented.

Hip-arthroplasty surgery and the inflammatory stress response in general affect the potential of recovery. Early postoperative orthostatic intolerance is common in patients undergoing THA with an incidence of 40%. The mechanism is thought related to an impaired autonomic regulation caused by surgery-induced inflammation. The effect of glucocorticoids on orthostatic intolerance, orthostatic hypotension and HRV after hip-arthroplasty surgery is unknown and calls for further investigation.

The study is to be considered as exploratory. The primary analysis of the primary outcome measure is a comparison of the incidence of orthostatic intolerance from baseline to 6 hours postoperatively between the two groups.

For calculation of sample size the difference in incidence between groups (40% versus 10%) from baseline (before surgery) to 6 hours after THA-surgery, a risk of type I errors 5% and a risk of type II errors 20% (80% power) were used.

The primary analysis is carried out on all included patients (intention-to-treat) with baseline values as covariate. Secondary exploratory per-protocol analysis might be performed. Missing outcomes will be analysed using multiple imputation due to expected strong time trends.

The secondary outcomes measures; Non-invasive blood pressure, systemic vascular resistance, cardiac output, HRV, plasma-hemoglobin, C-reactive protein.

For further details please also view the European Clinical Trials Database (EudraCT) registration:

EudraCT nr.: 2015-000102-19

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthrosis
* Undergoing total unilateral hip-arthroplasty surgery
* Speak and understand Danish
* Have given informed content

Exclusion Criteria:

* Revision or bilateral hip-arthroplasty surgery
* General anaesthesia
* Allergy or intolerance towards Methylprednisolone
* Local or systemic infection
* Permanent systemic treatment with steroids within 30 days peroperatively
* Insulin-dependent diabetes
* Atrial fibrillation
* Neurological disease incl. Parkinsons
* Daily use of hypnotics or sedatives
* Alcohol abuse >35 units per week
* Active treatment of ulcer within 3 months preoperatively
* Cancer disease
* Autoimmune disease incl. rheumatoid arthritis
* Pregnant or breast feeding women
* Menopause <1 year

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Difference in incidence of orthostatic intolerance from baseline to 6 hours after surgery | 6 hours after surgery

SECONDARY OUTCOMES:
Difference in incidence of orthostatic intolerance from baseline to 24 hours after surgery | 24 hours after surgery
Change in non-invasive blood pressure from baseline to 24 hours after surgery | 24 hours after surgery
Change in heart rate variability from baseline to 24 hours after surgery | 24 hours after surgery
Change in stroke volume and cardiac output from baseline to 24 hours after surgery | 24 hours after surgery
Change in systemic vascular resistance from baseline to 24 hours after surgery | 24 hours after surgery
Change in pain intensity from baseline to 24 hours after surgery | 24 hours after surgery
Change in concentration of plasma-hemoglobin from baseline to 48 hours after surgery | 48 hours after surgery
Change in concentration of C-reactive protein from baseline to 48 hours after surgery | 48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Viktoria Lindberg-Larsen, MD, Principal Investigator — Section for Surgical Pathophysiology, Rigshospitalet
Locations (1):
- Copenhagen University Hospital, Bispebjerg, Copenhagen NV, Denmark

REFERENCES:
- [Background] Husted H. Fast-track hip and knee arthroplasty: clinical and organizational aspects. Acta Orthop Suppl. 2012 Oct;83(346):1-39. doi: 10.3109/17453674.2012.700593. PMID 23205862
- [Background] Kehlet H. Fast-track hip and knee arthroplasty. Lancet. 2013 May 11;381(9878):1600-2. doi: 10.1016/S0140-6736(13)61003-X. No abstract available. PMID 23663938
- [Background] Grubb BP. Neurocardiogenic syncope and related disorders of orthostatic intolerance. Circulation. 2005 Jun 7;111(22):2997-3006. doi: 10.1161/CIRCULATIONAHA.104.482018. No abstract available. PMID 15939833
- [Background] Bundgaard-Nielsen M, Jans O, Muller RG, Korshin A, Ruhnau B, Bie P, Secher NH, Kehlet H. Does goal-directed fluid therapy affect postoperative orthostatic intolerance?: A randomized trial. Anesthesiology. 2013 Oct;119(4):813-23. doi: 10.1097/ALN.0b013e31829ce4ea. PMID 23756453
- [Background] Bundgaard-Nielsen M, Jorgensen CC, Jorgensen TB, Ruhnau B, Secher NH, Kehlet H. Orthostatic intolerance and the cardiovascular response to early postoperative mobilization. Br J Anaesth. 2009 Jun;102(6):756-62. doi: 10.1093/bja/aep083. Epub 2009 Apr 27. PMID 19398452
- [Result] Jans O, Bundgaard-Nielsen M, Solgaard S, Johansson PI, Kehlet H. Orthostatic intolerance during early mobilization after fast-track hip arthroplasty. Br J Anaesth. 2012 Mar;108(3):436-43. doi: 10.1093/bja/aer403. Epub 2011 Dec 15. PMID 22174345
- [Derived] Lindberg-Larsen V, Petersen PB, Jans O, Beck T, Kehlet H. Effect of pre-operative methylprednisolone on orthostatic hypotension during early mobilization after total hip arthroplasty. Acta Anaesthesiol Scand. 2018 Aug;62(7):882-892. doi: 10.1111/aas.13108. Epub 2018 Mar 24. PMID 29573263